CLINICAL TRIAL: NCT05063656
Title: Biomarker-Driven Pharmacological Treatment for Autism Spectrum Disorder
Brief Title: Biomarker-Driven Pharmacological Treatment of Adolescents With Autism Spectrum Disorder With Gabapentin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: David Cochran (Other)
Collaborators: Eagles Autism Foundation (Unknown)
Responsible Party: Sponsor-Investigator, David Cochran, Assistant Professor of Psychiatry and Pediatrics, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000151
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: social cognition; GABA; gabapentin; magnetic resonance spectroscopy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Open-label treatment with gabapentin for 8 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gabapentin Open-label treatment (Experimental): 8-week treatment with gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 8 weeks of gabapentin, titrated up to 20 mg/kg in 3 divided doses daily

SUMMARY:
The social cognitive deficits associated with autism spectrum disorder (ASD) are related to an imbalance in excitatory and inhibitory neurotransmission, specifically a deficit in the inhibitory neurotransmitter GABA. The investigators have used magnetic resonance spectroscopy (MRS) techniques to measure GABA in specific brain regions and have demonstrated that a single dose of gabapentin increases GABA in brain regions associated with social cognition. This study will use a biomarker-driven approach to investigate gabapentin to correct the underlying imbalance of neurotransmitters and improve the core social cognitive deficits in ASD. By using a brain-based biomarker (GABA) that is quantifiable and measurable, the investigators can target this biomarker directly and measure the impact of the treatment. This will help with the future development of targeted therapies for ASD and provide an early marker of response to aid in the selection of individuals more likely to respond to various treatments. The specific aims of this study are to: 1) determine if treatment with gabapentin sustainably increases GABA in the right anterior insula (RAI; an area of the brain involved in social cognition), 2) determine if response of RAI GABA levels to a single dose challenge of gabapentin predicts a sustained response after treatment, and 3) determine if the increase in GABA levels with gabapentin treatment translates into clinically measurable improvement in social cognition. The investigators will conduct an 8-week open-label clinical trial of gabapentin in 40 adolescents (age 13-17 years) with ASD, using MRS before and after treatment to measure GABA in the RAI (the primary outcome for the study). Before the trial, a single dose challenge of gabapentin will be used to evaluate the immediate response of GABA levels in the RAI, to determine if this predicts later response. A secondary outcome will be the clinical effects of gabapentin on social cognition. This study can demonstrate for the first time that neuroimaging biomarkers can be used to guide treatment of social cognition deficits seen in ASD and that the excitatory-inhibitory imbalance in neurotransmitters in ASD can be pharmacologically targeted. This can provide a rational basis for pharmacological treatment of the core social deficits of ASD, providing direct benefit to participants in the study as well as indirect benefit to countless patients in the future.

DETAILED DESCRIPTION:
1. Outline of Research Plan The investigators will recruit 40 adolescents with ASD (age 13-17) to participate in an 8-week open label clinical trial of gabapentin, with wraparound neuroimaging to assess the primary outcome of Aim 1 (response of RAI GABA levels to 8 weeks of gabapentin treatment) and Aim 2 (evaluation of acute response to gabapentin as a predictor of response at 8 weeks). Clinical measures of social cognition described below will be obtained to address Aim 3 (to assess for clinically measurable improvements in social cognition deficits).
2. Clinical Assessments The subjects will be assessed with the Autism Diagnostic Observation Schedule (ADOS-2) and Autism Diagnostic Interview-Revised (ADI-R) to confirm the diagnosis of ASD. The Ohio Autism Clinical Impressions Scale will assess overall severity of autism-specific symptoms. The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID 7.0.2) will be used to document comorbid psychiatric diagnoses. The Weschler Abbreviated Scales of Intelligence (WASI-2) will be used to assess IQ. Social cognition deficits will be assessed using the Reading the Mind in the Eyes test (RMET), the Social Responsiveness Scale (SRS-2), and the Vineland Adaptive Behavior Scales-II (VABS-II) Socialization subdomain. The Aberrant Behavior Checklist, Community version (ABC), will be used to quantify behavioral measures associated with ASD. To assess whether clinical improvements with gabapentin extend beyond effects on social cognition, other symptom domains will be assessed pre- and post-treatment as well. Specifically, information on repetitive and/or compulsive behaviors will be obtained using the Children's Yale-Brown Obsessive Compulsive Scale modified for Pervasive Developmental Disorders (CY-BOCS-PDD). The ADHD Rating Scale-IV (ADHD RS-IV) will be used to assess ADHD symptoms, the Children's Depression Rating Scale (CDRS) to assess depressive symptoms and the Multidimensional Anxiety Scale for Children, 2nd edition, (MASC-2) will be used to assess anxiety-related symptoms.

   In addition to traditional outcome measures for social functioning in ASD, including parent report measures (SRS-2) and theory of mind tasks (RMET), a novel technique of measuring social motor coordination will be used that was developed as a potential outcome measure in ASD clinical trials. This assessment involves a video-based analysis of whole-body social motor coordination during a more naturalistic task, the conversation task of an ADOS-2 administration. Changes in social motor coordination will be evaluated in relation to changes in GABA levels with treatment over the course of the clinical trial.
3. Baseline MRI T1- and T2-weighted high-resolution structural imaging (T1- and T2-weighted (MPRAGE)) will be acquired, along with a baseline MRS using MEsher-Garwood Point REsolved Spectroscopy Sequence (MEGA-PRESS: TE: 68 ms, TR: 2 s) to quantify GABA in a 4 cm x 2.5 cm x 2.5 cm voxel localized in the RAI. Imaging sessions will be conducted at the Advanced MRI Center (AMRIC) at UMMS, which houses a 3.0 Tesla Philips Achieva MRI research scanner (Philips Healthcare, Best, Netherlands) and 8 element phase-array receiver SENSE head coil.

   The baseline MRI protocol also leverages collaborations with the Human Connectome (HCP) and Adolescent Brain Cognitive Developments (ABCD) projects and is designed to support integration with national multi-site studies for added protocol utility. The scan session will include 1) a 3D T1-weighted magnetization-prepared rapid acquisition gradient echo scan for cortical and subcortical segmentation (6.5 min); 2) a 3D T2-weighted variable flip angle fast spin echo scan for screening out white matter lesions and quantification of CSF (6 min); 3) a diffusion imaging scan, for segmentation of white matter tracts and measurement of diffusion parameters (1.5mm isotropic, b=1000; 110 directions acquired with both AP and PA phase encoding; 2 x 5 min); 4) a resting state fMRI scan (2mm isotropic ; TR 750 ms; AP, PA phase encoding; (2-5.75 min runs).
4. Acute Response of GABA levels A second MRS scan will be obtained two hours after an approximately 20 mg/kg challenge with gabapentin to obtain the acute response for Aim 2. Subjects will receive a single dose of gabapentin. The dose used will be calculated to provide the highest possible dose to the nearest 100 mg without exceeding 1500 mg or 20 mg/kg, whichever is lower. The weight exclusion criteria ensures that all subjects will receive at least 17 mg/kg dose. All subjects will be monitored for adverse effects for up to 4 hours following administration of the single dose and will have direct phone access to the principal investigator (24 hours/ 7 days a week) for reporting of any post-observation adverse effects. A blood sample to assess drug level will be taken as close to 3 hours after administration as possible, allowing time for imaging scan and transport to clinical trials unit for blood draw. This will be used to control for variability in bioavailability in interpreting the cortical GABA level changes.
5. Clinical Trial of Gabapentin The study involves an 8-week open-label clinical trial with gabapentin in 40 adolescents age 13-17 years who meet DSM-5 criteria for ASD. At the acute gabapentin dosing visit, baseline safety labs will be obtained, including complete blood count; comprehensive metabolic panel including electrolytes, renal function tests, and liver function tests; and creatine kinase. Baseline EKG will be obtained as well. The above labs will be repeated at week 4 and week 8 of the clinical trial, or if adverse events occur which indicate the need for testing.

At baseline and at Weeks 2, 4, and 8, the following clinical measures will be obtained: OACIS-S, OACIS-I (for post-baseline visits). At baseline and at 8 weeks, the following assessments will also be administered: VABS-II, SRS-2 (modified to ask about symptoms in previous 2 weeks), RMET, ABC, CY-BOCS-PDD, ADHD-RS-IV, MASC-2, and CDRS-R. ADOS-2 will also be re-administered at week 8 for videotape assessment of social motor coordination as described above. At week 8, a trough serum gabapentin level will be obtained to account for variability in bioavailability as a potential confounding factor. At week 8, the MRS scan will be repeated to evaluate RAI GABA levels, and also include a resting state functional MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 years
* English as primary language (both child and legal guardian)
* DSM-5 criteria for Autism Spectrum Disorder
* IQ >70 per Weschler Abbreviated Scale of Intelligence (WASI)
* Informed assent for the study (The guardian must also give written informed consent)
* For sexually active females, agreement to use two forms of contraception during trial to avoid pregnancy

Exclusion Criteria:

* Any neurological disorder (e.g., cerebral palsy, fetal alcohol syndrome, cerebral neoplasm, bacterial meningitis, epilepsy, etc.)
* Genetic disorders (e.g., Fragile X, Rett Syndrome, etc.)
* Contraindications for MRI, such as metallic or electronic implants in the body, or severe claustrophobia
* Unstable psychiatric disorder expected to require psychotropic medication changes over the course of the study
* History of psychotic disorder
* Any condition that would prevent the subject from being able to complete study protocol
* Unstable medical illness such as diabetes, asthma, thyroid disease
* Currently on medications that cause respiratory depression, e.g. opioids, benzodiazepines
* Clinically significant suicidal ideation as assessed by the Columbia Suicide Severity Rating Scale
* History of intolerance to gabapentin or pregabalin
* Current substance use (including nicotine)
* Current treatment with gabapentin
* History of renal dysfunction
* Pregnancy in female participants.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Right Anterior Insula GABA level | 8 weeks
  Cortical GABA Levels in right anterior insula as measured by magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: David Cochran, MD, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication
Access Criteria: Available upon request from primary contact person